CLINICAL TRIAL: NCT01811186
Title: An Interventional Study to Compare the Efficacy and Tolerability of Current and Slow Titration With Targin® in the Treatment of Moderate to Severe Non-malignant Chronic Pain (GLORY)
Brief Title: An Interventional Study to Compare the Efficacy and Tolerability With Targin® in Non-malignant Chronic Pain (GLORY)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OXN12-KR-403
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Chronic Pain
Keywords: moderate to severe non-malignant chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Start oxycodone/naloxone 10/5mg b.i.d. titration->20/10mg b.i.d.->30/15mg b.i.d->40/20mg b.i.d.
  Interventions: Drug: Oxycodone/naloxone
- Group B (Other): Start oxycodone/naloxone 5/2.5mg b.i.d titration-> 10/5mg b.i.d.->20/10mg b.i.d.->30/15mg b.i.d->40/20mg b.i.d.
  Interventions: Drug: Oxycodone/naloxone

INTERVENTIONS:
Drug: Oxycodone/naloxone — Oxycodone/naloxone titration
  Other Names: Targin

SUMMARY:
Objectives:

1. Objective of main interest

   - To assess the drop-out rate caused by adverse event* after 6 weeks treatment
2. Further objectives

   * To assess the drop-out rate caused by adverse event* after 1 week treatment
   * To assess the pain reduction rate after 6 weeks treatment from baseline
   * To assess the Euroquol (EQ-5D) quality of life
   * To assess physician's overall satisfaction
   * To assess subject's overall satisfaction
   * To assess safety

DETAILED DESCRIPTION:
Study Design (Methodology):

This will be a single center, open-label, randomised, phase IV, exploratory interventional study to compare the efficacy and tolerability of current titration patterns and slow titration pattern with Targin® (Oxycodone/Naloxone) in the treatment of moderate to severe non-malignant chronic pain patients who are dissatisfied with their current analgesic medication World Health Organisation (WHO) step II analgesics).

Upon providing written informed consent, subject will be screened in the study and assessment will be performed at that time such as safety laboratory assessments, physical examination, vital sign, medical history taking, 24 hours pain intensity score. If the patient is eligible in inclusion/exclusion criteria at the time of visit 1, the patient will be randomized in a 1:1 ratio to allocate in Group A or Group B. Re-screening, study drug dose interruption is not allowed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 20 and <80 years of age
* Patients who have non-malignant chronic pain(≥90 days)
* Patients who have moderate to severe pain intensity which is not controlled with non-strong opioid
* Naïve patients for Oxycodone/Naloxone (Naïve patient defined as who did not treated for 90 days)
* Naïve patients for strong opioid (Naïve patient defined as who did not treated for 90 days)
* Patients who signed a written informed consent form

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
* Patients with known hypersensitivity to Oxycodone/Naloxone or to any of the excipients
* Patient who needs acute dose titration or whose pain intensity fluctuate significantly in a short period according to investigator's judgment
* Having used other investigational drugs at the time of enrollment, or within 30 days of enrollment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoseong Lee, Dr., Principal Investigator — Asan Medical Center
Locations (1):
- AMC, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety set: 261 patients were enrolled. ITT set was 258, 3 patients of the 261 patients deviated from inclusion/exclusion criteria.
Groups:
- Start Oxycodone/Naloxone 10/5mg b.i.d.: Start oxycodone/naloxone 10/5mg b.i.d. titration->20/10mg b.i.d.->30/15mg b.i.d->40/20mg b.i.d.
- Start Oxycodone/Naloxone 5/2.5mg b.i.d: Start oxycodone/naloxone 5/2.5mg b.i.d->10/5mg b.i.d. titration->20/10mg b.i.d.->30/15mg b.i.d->40/20mg b.i.d.
Period: Overall Study
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d. | Start Oxycodone/Naloxone 5/2.5mg b.i.d
Started | 132 | 126
Completed | 61 | 64
Not Completed | 71 | 62
Not completed — Adverse Event | 54 | 38
Not completed — Protocol Violation | 5 | 6
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Lack of Efficacy | 3 | 6
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety set: 261 ITT set: 258(3 patients were deviated inclusion/exclusion criteria among 261)
Groups:
- Start Oxycodone/Naloxone 5/2.5mg b.i.d: Start oxycodone/naloxone 5/2.5mg b.i.d titration-> 10/5mg b.i.d.->20/10mg b.i.d.->30/15mg b.i.d->40/20mg b.i.d.
- Total: Total of all reporting groups
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d | Start Oxycodone/Naloxone 5/2.5mg b.i.d | Total
Number analyzed (Participants) | 132 | 126 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 64 | 141
  >=65 years | 55 | 62 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.63 (9.69) | 61.15 (11.94) | 60.88 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 84 | 165
  Male | 51 | 42 | 93
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 132 | 126 | 258

OUTCOME MEASURES:

1. Primary Outcome: Drop-out Rate Caused by Adverse Event After 6 Weeks Treatment
Description: To assess the drop-out rate caused by adverse event* after 6 weeks treatment
Time Frame: 6 weeks
Population: Intent to treat analysis set: 258 patients (Last Observation Carried Forward)
Measure: Number; unit: percentage of participants
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d. | Start Oxycodone/Naloxone 5/2.5mg b.i.d.
Number analyzed (Participants) | 132 | 126
percentage of participants | 40.91 | 30.16

2. Secondary Outcome: The Drop-out Rate Due to an Adverse Event After 1 Week Treatment With the Study Drug.
Description: The drop-out rate due to an adverse event after treatment (1 week) by treatment arm were summarized and presented as frequency and percentage, and the inter-group difference were compared by using a Chi-square test or Fisher's exact test.
Time Frame: 1 week
Population: Intent to treat analysis set: 258(Last observation Carried Forward)
Measure: Number; unit: percentage of participants
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d. | Start Oxycodone/Naloxone 5/2.5mg b.i.d.
Number analyzed (Participants) | 132 | 126
percentage of participants | 28.79 | 19.84

3. Secondary Outcome: The Change of Pain Intensity Scores(NRS) From Baseline After 6 Weeks Treatment With the Study.
Description: Change in numeric rating scales (NRS) such as score for average pain levels over the previous 24 hours, from baseline to 6weeks. NRS score was measured from 0 (No pain) to 10(worst pain imaginable).
Time Frame: 6 weeks
Population: ITT analysis set: 258
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d. | Start Oxycodone/Naloxone 5/2.5mg b.i.d.
Number analyzed (Participants) | 132 | 126
units on a scale | -1.62 (1.90) | -1.48 (1.82)

4. Secondary Outcome: Change of Quality of Life (EQ-5D) Score After 6 Weeks Treatment With the Study Drug
Description: EQ-5D to measure of health related quality of life should be answered as one of 3 levels about current condition for 5 dimensions and was calculated total average by giving a weighting on 3 level of answers (EQ-5D levels into 'no problems' (level 1) and 'problems' (level 2 and 3)).
  Table of scores by each level for EQ-5D items: mobility(level 1=0, level2=0.069,level 3=0.314), self care(level 1=0, level2=0.104,level 3=0.214), usual activities(level 1=0, level2=0.036,level 3=0.094), pain/discomfort (level 1=0, level2=0.,level 3=0.386) and anxiety/depression(level 1=0, level2=0.071,level 3=0.2)
  *EQ-5D Total = 1 - 0.081 - (the score of the each level) - 0.269 (if at least one of level 3 presents)
  EQ-5D total score could be 0.919 in maximum and -0.594 in minimum if case all index indicates the level 3. So, if EQ-5D total score closed by "1" means that the healthy condition and high quality of life.
Time Frame: 6 weeks
Population: ITT analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d. | Start Oxycodone/Naloxone 5/2.5mg b.i.d.
Number analyzed (Participants) | 61 | 64
units on a scale | 0.14 (0.26) | 0.07 (0.22)

5. Secondary Outcome: Assessment of Investigator's Overall Satisfaction After 6 Weeks Treatment With the Study Drug
Description: Investigator's overall satisfaction after treatment (6 weeks) (Clinical Global Impression of Change Scale(CGIC) 7 point scale) by treatment arm were summarized and presented as frequency and proportion, and the inter-group difference were compared by using a Chi-square test or Fisher's exact test.
Time Frame: 6 weeks
Population: ITT analysis set: 171. Last visit(Visit 5) data was handled as LOCF. However, Missing Number as visit 3 for assessment of Investigator's overall satisfaction after 6 weeks treatment with the study drug was Group A = 50, Group B=37.
Measure: Number; unit: participants
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d | Start Oxycodone/Naloxone 5/2.5mg b.i.d
Number analyzed (Participants) | 82 | 89
participants
  Very much improved | 2 | 2
  Much improved | 27 | 30
  Minimally improved | 48 | 43
  No change | 5 | 14
  Minimally worse | 0 | 0
  Much worse | 0 | 0
  very much worse | 0 | 0

6. Secondary Outcome: Assessment of Subject's Overall Satisfaction After 6 Weeks Treatment With the Study Drug
Description: At each visit, the subject assessed the overall satisfaction for efficacy by using the 7 point scale of Patient Global Impression of Change Scale(PGIC).
Time Frame: 6weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d. | Start Oxycodone/Naloxone 5/2.5mg b.i.d.
Number analyzed (Participants) | 82 | 89
participants
  Very much improved | 2 | 2
  Much improved | 24 | 28
  Minimally improved | 44 | 42
  No change | 11 | 16
  Minimally worse | 0 | 1
  Much worse | 1 | 0
  Very much worse | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety set: Safety set included data obtained from all subjects who administered at least one dose of the study drug. Patients were followed by 6 weeks.
Arm/Group | Start Oxycodone/Naloxone 10/5mg b.i.d | Start Oxycodone/Naloxone 5/2.5mg b.i.d
Serious Adverse Events (participants affected / at risk) | 0/133 | 2/128
Other Adverse Events (participants affected / at risk) | 115/133 | 104/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Start Oxycodone/Naloxone 10/5mg b.i.d (N=133) | Start Oxycodone/Naloxone 5/2.5mg b.i.d (N=128)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) — They all resolved during the study and they were all evaluated as 'Unrelated' to the study drug.
Inflammation (General disorders) | 0 (0) | 1 (1) — system organ class: General disorders and administration site conditions
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Start Oxycodone/Naloxone 10/5mg b.i.d (N=133) | Start Oxycodone/Naloxone 5/2.5mg b.i.d (N=128)
Nausea (Gastrointestinal disorders) | 52 (55) | 46 (53)
Constipation (Gastrointestinal disorders) | 24 (26) | 21 (21)
vomiting (Gastrointestinal disorders) | 27 (27) | 16 (16)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 32 (34) | 29 (29)
Somnolence (Nervous system disorders) | 21 (22) | 26 (27)
Headache (Nervous system disorders) | 15 (16) | 8 (10)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Mental impairment (Nervous system disorders) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (21) | 17 (17)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 4 (4)
Oedema (General disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Dysuria (Renal and urinary disorders) | 4 (4) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No